CLINICAL TRIAL: NCT04861038
Title: Study Using Negative Pressure to Reduce Apnea (SUPRA)
Brief Title: Study Using Negative Pressure to Reduce Apnea
Acronym: SUPRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sommetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOM-029
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Sleep Apnea, Obstructive; Apnea, Sleep
Keywords: sleep apnea; OSA; obstructive sleep apnea; CPAP failure; apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- aerSleep II (Experimental): Use of aerSleep II device to provide continuous external negative pressure to treat moderate to severe OSA in spontaneously breathing subjects who are intolerant of CPAP
  Interventions: Device: aerSleep II

INTERVENTIONS:
Device: aerSleep II — Continuous negative external pressure (cNEP) system that maintains an open airway by applying negative pressure to the anterior neck via a soft silicone collar

SUMMARY:
The objective of this study is to determine the safety and effectiveness of the aerSleep® II device for treatment of moderate to severe Obstructive Sleep Apnea (OSA) over 24 weeks of home use in spontaneously breathing adult subjects who are intolerant of Continuous Positive Airway Pressure (CPAP) therapy.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, prospective, observational intervention study to determine the safety and effectiveness of the aerSleep II System. Up to 900 subjects will be enrolled at up to 30 study sites in the United States and outside the United States to ensure that approximately 79 subjects who are termed initial responders can be evaluated after 24 weeks of home use with the aerSleep II device. As part of screening and prior to intervention, home sleep testing will be performed to establish baseline apnea-hypopnea index (AHI). Subjects meeting study criteria will wear the aerSleep II device at home. After a 1-week period of acclimation, subjects will have a second HST (HST #2). Initial responders with a ≥50% reduction in AHI from baseline with an AHI <20/hour will be continued on home treatment. Non-responders will be discontinued from the study. After 12 weeks, subjects will have an interim home sleep study. After 24 weeks of home use, subjects will have HST #4 to determine the primary effectiveness endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Body mass index ≤42 kg/m2
3. Prior documented diagnosis of OSA by means of a polysomnography (PSG) test or home sleep test (HST)
4. Documented evidence from a screening HST following consent to demonstrate:

   1. AHI 15 - 50/hour
   2. >80% of the apneas and hypopneas are obstructive
5. Previous treatment attempt with CPAP resulting in failure to treat or discontinuation due to intolerance, subject choice, or struggle to use CPAP
6. Have not used CPAP or oral appliances within 1 week of the screening home sleep test and agree not to use CPAP or oral appliances throughout the study duration
7. Access to and ability to use a smart device such as a smartphone or tablet
8. Able to speak, read, and write English
9. In the opinion of the investigator, the subject will be able to understand and comply with all study procedures.

Exclusion Criteria:

1. Known sleep disorder other than OSA, such as narcolepsy, restless leg syndrome, idiopathic hypersomnolence or chronic insomnia
2. Craniofacial abnormalities that may be contributing to OSA
3. Previous surgery, injury, or radiation to the neck which, in the Investigator's judgment, could interfere with collar fit or comfort
4. Excessive hair or beard in the area of the neck where the collar will be placed, and/or unwillingness to shave that area for the duration of this study
5. Inflammatory skin condition, such as acne or eczema in the area where the collar will be affixed to the skin, which, in the Investigator's judgment, could interfere with collar fit or comfort
6. Known silicone allergy
7. Night shift work because of irregular sleep-wake cycles
8. Excessive alcohol intake, defined as that leading to interference with work, home life, or the ability to optimally perform normal everyday duties and tasks
9. Use of illicit drugs currently or within the past 5 years
10. Serious pulmonary disease (e.g., cor pulmonale, CO2 retention, or poorly controlled asthma)
11. Use of home oxygen or baseline oxygen saturation <94%
12. Cancer that has been in remission for less than one year
13. Psychiatric illness that, in the opinion of the Investigator, is not reasonably well-controlled with treatment
14. Serious cardiac disease (e.g., congestive heart failure, unstable coronary artery disease, or poorly controlled rhythm disturbance)
15. Prior carotid endarterectomy, prior percutaneous coronary angiography (including any placement of carotid stents), or known stenosis of either internal carotid artery > 70% from prior carotid imaging (e.g., carotid duplex ultrasound, angiography, computed tomography angiography, or magnetic resonance angiography)
16. Previous surgery for peripheral arterial disease
17. Presence of possible or definite carotid artery disease, defined as any of the following:

    1. history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) with uncertain etiology that is compatible with carotid artery disease
    2. diminished carotid pulse on screening physical examination*
    3. > 70% stenosis in either extra-cranial internal carotid artery as determined by duplex ultrasound* (only performed on those who do not exhibit 17 a. or b.)
18. Tonsil size 3 or 4 (Appendix C)*
19. Currently pregnant* or planning to become pregnant during participation in this study
20. Unable to obtain adequate collar fit*
21. Any condition or circumstance that, in the opinion of the investigator, may preclude study completion, interfere with accurate data collection, or bias the results
22. The investigator believes that the subject's participation may not be in his or her best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sustained response to aerSleep II therapy at 24 weeks | 24 weeks
  The primary effectiveness endpoint is to demonstrate that a majority of adult subjects who are initial responders to aerSleep II therapy experience a change of at least 50% of their baseline AHI with an AHI rate less than 20 per hour at the final home sleep test at 24 weeks.
Adverse Device Effects | 24 weeks
  The primary safety endpoint is to characterize the adverse device effects experienced throughout the study.

SECONDARY OUTCOMES:
ODI change | 24 weeks
  Demonstrate a change in Oxygen Desaturation Index (ODI) at HST #4 compared to baseline HST for initial responders
AHI change from baseline for all subjects that acclimate to the aerSleep II device | 24 weeks
  Determine the proportion of subjects that acclimate to the device that exhibit a change in AHI after 24 weeks of home use with the aerSleep II device
Change in sleep disturbance from baseline as measured by Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance questionnaire | 24 weeks
  Determine the change in sleep disturbance at the end of the study compared to baseline using the validated PROMIS Short Form Sleep Disturbance 8b questionnaire
Change in sleep impairment from baseline as measured by PROMIS Sleep Sleep-Related Impairment questionnaire | 24 weeks
  Determine the change in sleep impairment at the end of the study from baseline as measured by the validated PROMIS Short Form Sleep-Related Impairment 8a questionnaire
Change in sleep from baseline as measured by Patient Global Impression Scale questionnaire | 24 weeks
  Determine any change in sleep at the end of the study from baseline as measured by the Patient Global Impression Scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kingman P. Strohl, M.D., Principal Investigator — Case Western Reserve University School of Medicine
Locations (15):
- United States (15):
  - University of Arizona, Tucson, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Infinitive Bioresearch, Los Angeles, California
  - BetterNight, San Diego, California
  - Delta Waves, Colorado Springs, Colorado
  - Baptist Hospital, Miami, Florida
  - Clayton Sleep Institute, St Louis, Missouri
  - The MetroHealth System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Bogan Sleep Consultants, Columbia, South Carolina
  - BioSerenity, Columbia, South Carolina
  - Sleep Therapy & Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No